CLINICAL TRIAL: NCT02976675
Title: Pegylated Somatropin (PEG Somatropin) in the Treatment of Children With Growth Hormone Deficiency: A Multicenter, Randomized, Open-label, Parallel Phase IV Clinical Trial With Different Administration Frequency of PEG Somatropin
Brief Title: Pegylated Somatropin (PEG Somatropin) in the Treatment of Children With Growth Hormone Deficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Children's Hospital of Fudan University (Other); Suzhou Municipal Hospital (Other); General Hospital of Ningxia Medical University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); Maternal and Child Health Hospital of Hubei Province (Other); Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 004 CT-4
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2016-11

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG-somatropin (Experimental): Pegylated somatropin, injection, 54IU/9.0mg/1.0ml/kit Group of dosing per week:0.20 mg /kg/w, once per week for 26 weeks
  Interventions: Biological: PEG-somatropin
- PEG-somatropin per two weeks (Experimental): Pegylated somatropin, injection, 54IU/9.0mg/1.0ml/kit Group of dosing per two weeks:0.20 mg /kg/2w，once per two weeks for 26 weeks
  Interventions: Biological: PEG-somatropin
- Jintropin AQ (Active Comparator): Jintropin AQ, injection, 30IU/10 mg/3ml/cartridge, 0.25mg/kg/w, once per day for 26 weeks
  Interventions: Biological: PEG-somatropin

INTERVENTIONS:
Biological: PEG-somatropin — Pegylated somatropin, injection, 54IU/9.0mg/1.0ml/bottle Group of dosing per week:0.20 mg /kg/w, once per week for 26 weeks
Biological: PEG-somatropin — Pegylated somatropin, injection, 54IU/9.0mg/1.0ml/bottle Group of dosing per two weeks:0.20 mg /kg/2w，once per two weeks for 26 weeks

SUMMARY:
To evaluate the safety and efficacy of PEG Somatropin Injection in the treatment of children with growth hormone deficiency, as well as to study the feasibility of extending the dosing intervals (once per two weeks) of PEG Somatropin Injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are diagnosed as GHD before starting treatment, according to medical history, clinical symptoms and signs, GH provocation tests and imaging and other examinations:

  1. According to statistical height data of physical development of Chinese children in nine cities in 2005, the height is lower than 3rd percentile growth curve of the same age, same sex normal children;
  2. Height velocity (HV) ≤5.0 cm / yr;
  3. GH provocative tests (with two drugs of different mechanism of action) confirmed plasma GH peak <10.0 ng / ml;
  4. bone age for girl≤9 years old, for Boy≤10 years old, bone age is one year or more later than the actual age, that is the actual age - bone age ≥ 1 year;
* Before puberty (Tanner I stage), age≥3 years old, male or female;
* Subjects have not received hormone therapy within 6 months;
* Subjects is willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures, to sign informed consent.

Exclusion Criteria:

* Dysfunction of liver and kidney (ALT> 2 times the upper limit of normal, Cr> upper limit of normal);
* Patients positive for hepatitis B c-antibody (HBcAb), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg);
* Patients with known hypersensitivity to PEG Somatropin or Somatropin or any other components of the study product;
* Patients with severe cardiopulmonary or hematological diseases, a current or past history of malignant tumors, immunodeficiency diseases, or mental diseases;
* Potential cancer patients (family history);
* Patients with diabetics;
* Patients with other growth disorders, such as Turner's syndrome, sexual physical delayed puberty, Laron syndrome, growth hormone receptor deficiency, girls with slowly growing who did not rule out chromosomal abnormalities;
* Patients with congenital bone dysplasia or scoliosis;
* Subjects took part in other clinical trial study during 3 months;
* Other conditions in which the investigator preclude enrollment into the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Ht SDSca | Baseline, 4,12,26 weeks after initiating treatment
  Ht SDSca was calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age

SECONDARY OUTCOMES:
Ht SDSBA | Baseline, 4,12,26 weeks after initiating treatment
  Calculate by formula
Yearly growth velocity | Baseline, 4,12,26 weeks after initiating treatment
  Calculate by formula
IGF-1SDS | Baseline, 4,12,26 weeks after initiating treatment
  Calculate by formula
IGF-1/IGFBP-3 molar ratio | Baseline, 4,12,26 weeks after initiating treatment
  Calculate by formula
Bone age | Baseline, 4,12,26 weeks after initiating treatment
  Calculate by formula

CONTACTS AND LOCATIONS:
Overall Officials: Feihong Luo, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (24):
- China (24):
  - Maternal and Child Health Hospital of Anhui province, Hefei, Anhui
  - First People's Hospital of Lu'an City, Lu'an, Anhui
  - Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Maternal and Child Health Hospital of Guiyang City, Guiyangtou, Guizhou
  - Maternal and Child Health Hospital of Hainan province, Haikou, Hainan
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - Maternal and Child Health Hospital of Hubei province, Wuhan, Hubei
  - First People's Hospital of Changzhou City, Changzhou, Jiangsu
  - First People's Hospital of Lianyungang City, Lianyungang, Jiangsu
  - Jiangsu Provincial Hospital of Chinese Traditional medicine, Nanjingkou, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Suzhou City Hospital, Suzhou, Jiangsu
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Maternal and Child Health Hospital of Tai'an city, Tai’an, Shandong
  - Children's Hospital of Chengdu city, Chengdu, Sichuan
  - People's Hospital of Cixi City, Cixi, Zhejiang
  - First People's Hospital, Hangzhou, Zhejiang
  - First People's Hospital of Jiaxing City, Jiaxing, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Jishuitan Hospital of Beijing City, Beijing
  - Peoples' hospital of Inner Mongolia Autonomous Region, Inner Mongolia Autonomous Region
  - General Hospital of Ningxia Medical University, Ningxia Autonomous Region
  - Children's Hospital of Fudan University, Shanghai

REFERENCES:
- [Derived] Sun C, Lu B, Liu Y, Zhang Y, Wei H, Hu X, Hu P, Zhao Q, Liu Y, Ye K, Wang K, Gu Z, Liu Z, Ye J, Zhang H, Zhu H, Jiang Z, Liu Y, Wan N, Yan C, Yin J, Ying L, Huang F, Yin Q, Xi L, Luo F, Cheng R. Reduced Effectiveness and Comparable Safety in Biweekly vs. Weekly PEGylated Recombinant Human Growth Hormone for Children With Growth Hormone Deficiency: A Phase IV Non-Inferiority Threshold Targeted Trial. Front Endocrinol (Lausanne). 2021 Nov 25;12:779365. doi: 10.3389/fendo.2021.779365. eCollection 2021. PMID 34899612